CLINICAL TRIAL: NCT06749002
Title: Additional Effects of Functional Muscle Training With Turning Based Specific Training During Turning in Post Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/61
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Subacute Stroke; Chronic Stroke; Balance
Keywords: Stroke; chronic stroke; functional muscle training; Turning based specific training; Turning in Gait
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): It includes participants receiving Functional muscle training along with Turning based specific training over a period of 6 weeks.
  Interventions: Procedure: Turning based specific training along with functional Muscle training
- Control Group (Active Comparator): It includes participants recieving Turning based specific training only for 6 weeks.
  Interventions: Procedure: turning based specific training.

INTERVENTIONS:
Procedure: Turning based specific training along with functional Muscle training — Experimental group will receive Turning based specific training protocol for 6 weeks along with functional muscle training, training will be done on alternate days.
  Functional muscle training:
  Details: Week 1-6: 3 days a week on alternate days.
  Hip Abductors:
  Side lying leg raises Single leg squatting Standing leg wall press Progressing to Adding resistance bands
  Hip adductors:
  Side lying adduction Standing Adduction Progress to adding resistance bands
  Hip Flexors:
  Standing leg lift Straight leg raises Progress to adding resistance bands
  Hip Extensors:
  Prone lying raises Standing single leg extension Progress to adding resistance bands
  Plantarflexors/ DorsiFlexors:
  Plantarflexors:
  Plantarflexion against resistance Toe raises
  Dorsiflexors:
  Dorsiflexion against resistance Heel raises
  Hip external rotators:
  Sitting-externally rotate hip 0-30° Add resistance bands
  Hip Internal rotators:
  Sitting-internally rotate the hip 0-30° Add resistance bands.
  Arms: Experimental group
Procedure: turning based specific training. — Week 1:
  90 Degrees turns on the spot
  Visual cues to follow
  Week 2-3:
  90 degrees turns on the spot
  Figure of 8 walking
  Visual cues to follow
  Week 4-5:
  90 Degrees turns on the spot
  Figure of 8 walking
  Step across body
  Braiding
  Week 6:
  90 degree turns on the spot
  Figure of 8 walking
  Step across body
  Braiding
  Visual cues to follow
  Obstacle avoidance
  Arms: Control Group

SUMMARY:
Stroke is the leading cause of disability leading to Gait and balance dysfunction leading to decreased Quality of Life. Difficulty in turning is a major target in Gait Rehabilitation. Task specific exercises has proven to be effective in all stages of stroke rehabilitation, therefore Turning based specific training is to be used in order to improve turning and balance in post stroke patients moreover functional strength training of lower extremities prove to be more effective than traditional training.

DETAILED DESCRIPTION:
The objectives of this study are:

1. To determine the additional effects of functional muscle training with turning based specific training on turning in Gait among post stroke patients.
2. To the determine the additional effects of functional muscle training with turning based specific training on balance in post stroke patients.
3. To determine the additional effects of functional muscle training with turning based specific training on Quality of LIfe aming post stroke patients.

HYPOTHESIS:

Alternate hypothesis 1.1HA-There will be a statistically significant difference of muscle training in addition with turning based specific training in turning among post stroke patients (p<0.05).

2. 2HA- There will be statistically significant difference between muscle training in addition with turning based specific training on balance in post stroke patients (p<0.05).

Null hypothesis:

1.1H0 -There will be statistically no significant difference of muscle training with turning based specific training on turning in Gait among post-stroke patients (p>0.05) 2 .2HO-There will be statistically no significant difference of muscle training with turning specific training on balance in post stroke patients (p>0.05)Research Design: Experimental study. Randomized Control Trial

Clinical setting: Rehabilitation department, Fauji Foundation Hospital.

Selection Criteria:

Inclusion Criteria

* Age group: 45-60 years onwards
* Both males and females
* Patients with subacute and chronic stroke (MCA >6months)
* MMSE- 25 or higher, Functional ambulatory capacity-3

Exclusion Criteria

* Hemorrhagic stroke.
* Patients with epilepsy
* Patients with other neurological conditions loke Alzheimer, parkinsons and dementias.

Sampling technique: non-probability purposive sampling.

Outcome Measures:

TURNING: 1) Standing Turn Test, 2) Figure of 8 Test. BALANCE: 1) Berg Balance Scale, 2) Timed up and Go Test, 3) Modified 4 square step Test.

Outcome measures will be evaluated at baseline and then after 6 weeks of intervention.

Experimental Group (A) = This group will recieve Turning based specific training along with Functional muscle training for 6 weeks.

Control group (B) = This group will recieive Turning Based Specific Training only for 6 weeks

Data analysis techniques:

The data will be analyzed through SPSS 21 and Data would be analyzed based on the study design chosen that is random control experimental study.

Significance of the study:

Turning is a major component of ambulation. Difficulty in turning results in increased risk of fall. Stroke results in step asymmetry which increases difficulty in changing direction.

There is sufficient evidence available for normal gait training but limited protocols for targetting turning in Gait.

The current study aims to fill this gap by providing research data and developing a treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age group: 45-60 years onwards
* Both males and females
* Subacute and chronic stroke (MCA >6months)
* MMSE score 25 or higher.
* FAC -3

Exclusion Criteria:

* Hemorrhagic stroke.
* Patients with Epilepsy.
* Patients with other neurological conditions like Alzheimer, Parkinson and other Dementias.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Turning performance. | 6 weeks
  Standing turn test will be used for turning performance
turning ability | 6 weeks
  Figure of 8 test will be used for turning ability
Balance | 6 weeks
  Berg Balance Scale will be used to assess balance
Balance | 6 weeks
  Four square stand test will be used for this

SECONDARY OUTCOMES:
Balance | 6 weeks
  Timed up and go test will be used for this

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Punjab Province, Pakistan